CLINICAL TRIAL: NCT05657730
Title: Analysis of the Intestinal Flora Composition After Consumption of Water Kefir
Brief Title: Study the Effect of Water Kefir Consumption on the Gut Microbiome in Healthy Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Åsa Håkansson, Associate Professor, Lund University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Water Kefir
Record Dates: First submitted 2022-11-09; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Healthy Diet; Gastrointestinal Microbiome; Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active group (Experimental)
  Interventions: Dietary Supplement: Water Kefir beverage

INTERVENTIONS:
Dietary Supplement: Water Kefir beverage — Participants will consume the water kefir beverage for two weeks.

SUMMARY:
The goal of this intervention study is to analyse the microbiota composition after the water kefir consumption. The main questions are to evaluate the potential probiotic drink can have beneficial effect on the gut microbiota. Participants will consume the water kefir for two weeks and microbiota will be analysed. Researchers will compare the microbiota composition before and after consumption.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age.
* must be able to complete the form digitally.

Exclusion Criteria:

* must not be diagnosed with gastrointestinal diseases, autoimmune diseases or have diseases or medications that cause immune deficiency such as MS, type 1 diabetes, cancer or HIV.
* must not take antibiotics during the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-01-14 (Estimated); Study Completion 2023-04-14 (Estimated)

PRIMARY OUTCOMES:
16S metagenomics based measurement of the bacterial diversity (alpha- and beta diversity indices), and the composition (relative abundance of the bacterial taxa in each sample) | up to 24 weeks
  Potential changes of microbiome after consumption of the water kefir will be assessed by analyzing the 16S metagenomics

CONTACTS AND LOCATIONS:
Locations (1):
- Lund University, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No